CLINICAL TRIAL: NCT06159569
Title: Open Not Comparative Clinical Trial on the Performance and Tolerability of the Medical Device LACRIACT, Eye Drops for the Treatment of Dry Eye
Brief Title: Performance and Tolerability of the Medical Device LACRIACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laboratórios Baldacci S.A (Industry)
Collaborators: Opera CRO, a TIGERMED Group Company (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LACRIACT 1/2020
Record Dates: First submitted 2023-11-28; First posted 2023-12-06 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Dry Eye; Contact Lens Acute Red Eye; Photophobia; Discomfort
Keywords: LACRIACT; Contact lens; Photophobia; Stickiness of eyelashes; Italy
MeSH Terms: conditions — Dry Eye Syndromes; Photophobia

STUDY DESIGN:
Intervention Model Description: Open, non comparative study with a medical device
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Population treated with LACRIACT (Experimental): 20 patients affected by dry eye who met the inclusion and exclusion criteria.. It is optional for the Investigator to recruit a sub-group of patients (maximum number 10 of 20 recruited patients) with regular soft contact lens that will be analysed separately.
  Interventions: Device: LACRIACT

INTERVENTIONS:
Device: LACRIACT — LACRIACT is is a preservative free ophthalmic sterile medical device solution. The solution is packaged in closable vials of inert material that does not affect the contents (clear low-density polyethylene), each vial contains 0.5 ml of solution.
  Eligible patients will start the treatment. Patients will receive the box of eye drops, and will be instructed on how to self-administer 1 drop in each eye 4 times a day for 30 days starting from the day following the visit.

SUMMARY:
The goal of this study is testing LACRIACT® eye drops, a medical device, to see how well it works and if people can use it safely. The Investigators will study this in people who have dry eyes, some of whom wear contact lenses, and some who do not. To obtain data from 20 participants, the investigators will first screen 22 patients, as two of them may not meet the requirements. If someone quits the study, the Investigators will not replace them with someone else.

A person can partecipate in the study if they meet certain criteria in the study plan, complete the entire treatment, and use eye drops correctly at least 80% of the time. The Investigators running the study might also include up to 10 people who wear soft contact lenses out of the 20 in total.

This study will be conducted at a clinic in Italy.

DETAILED DESCRIPTION:
Dry eye disease is defined as a multifactorial disease of the tears and ocular surface that results in symptoms of discomfort, visual disturbance, and tear film instability with potential damage to the ocular surface. It is accompanied by increased osmolarity of the tear film and subacute inflammation of the ocular surface (Ocul Surf. 2007;5(2):75). Tear hyperosmolarity is responsible for several morphological changes in conjunctival and corneal cells, and stimulation of the inflammatory cascade, resulting in the release of mediators such as cytokines and proteolytic enzymes, loss of both mucin-producing goblet cells and corneal barrier function. The international literature shows that ophthalmic products containing the biologic glycosaminoglycan sodium hyaluronate (HA) at concentrations around 0.2% (between 0.15% and 0.25%) are well tolerated and no safety problems have been reported. In fact, being hydrophilic, HA binds a large amount of water and forms a viscous hydrated gel even at low concentrations, which helps to restore and stabilize the compromised tear film in dry eye patients. Recently, the use of osmoprotectants, which are able to counteract the hyperosmolarity of the tear film, has been evaluated as a beneficial strategy for the treatment of dry eye. Osmoprotection can be considered as a natural response of biological structures that, through the accumulation of small biological molecules on cell surfaces, causes an adaptation of these structures to a hyperosmotic environment. For this reason, the selection of new osmoprotective agents for the treatment of dry eye should be a goal of current clinical research in ophthalmology. LABORATORI BALDACCI has recently selected 5-oxo-2-pyrrolidinecarboxylic acid (PCA), known as pyroglutamic acid, an endogenous molecule able to meet the expectations of demonstrating beneficial behavior in reducing dry eye symptoms. The medical literature (Tampucci S et al, Pharmaceutics. 2018), demonstrated that the scarce tear volume in contact with the corneal epithelial cells in atropine-induced dry eye in rabbits was influenced by the presence of hydrophilic PCA, which was able to provide protection against desiccation due to its osmoprotective activity and high water-binding capacity, thereby maintaining a significant tear volume in the conjunctival sac. Furthermore, the combination of PCA and HA allows for a significant improvement in this behavior, probably due to the ability of HA to hold approximately 1000 times its weight in water with respect to the surrounding tissue. These positive preclinical results should be confirmed in the ongoing clinical trials. The combination of PCA as an osmoprotective agent and HA as a pharmaceutical mucoadhesive and viscosifying agent capable of optimizing the ocular pharmacokinetic behavior of PCA may be a promising combination for the treatment of dry eye.

LACRIACT®, the medical device ophthalmic solution used in this clinical trial, was designed to act locally without the need for systemic absorption. In fact, PCA and HA are physiological substances that do not present toxicity issues. LACRIACT® was formulated to alleviate dry eye symptoms through localized physical action, without involvement of any immunological or pharmacological activity, and minimizing discomfort upon application.

This open, non-randomized trial will take place at an Italian clinical site. The purpose is to assess the performance, safety, and tolerability of LACRIACT® eye drops in patients with mild to moderate dry eye syndrome, with or without contact lenses. The investigators opted to treat solely mild to moderate dry eye because severe forms of dry eye necessitate a comprehensive approach where tear substitutes constitute only a part of the therapy. Assessing the efficacy and tolerance of LACRIACT becomes more complex when used with concomitant local and systemic dry eye treatments. The sample size has been determined to be 20 evaluable patients, and the Investigators plan to screen 22 patients to achieve this number (allowing for 2 screening failures). Dropouts will not be replaced. The Investigator may include a maximum of 10 patients (out of a total of 20) who regularly wear soft contact lenses, but this is optional.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both genders aged 18-75;
* Patients with clinically diagnosed mild to moderate dry eye syndrome based on Ocular Surface Disesae Index OSDI questionnaire (Italian version) and medical examination;
* Patients with at least two signs and/or symptoms of ocular discomfort;
* Patients with good eyelid mobility;
* Patients must be able to attend the visits scheduled in the study protocol and to follow the instructions given by the Investigator;
* Patients must be able to fill in their diary at home;
* Patients who have given their written informed consent.

Exclusion Criteria:

* Ocular hypertension (>21 mmHg) or glaucoma with/without alterations of the field of vision;
* Presence of any other eye acute conditions different from eye dry (e.g. acute ulcerative keratitis; acute purulent ophthalmia; ocular tuberculosis; ocular mycosis);
* Eye inflammation or acute eye infection within 3 months before the enrolment;
* Eye surgery within 1 year before enrolment or LASIK at any time before enrolment;
* Known hypersensitivity to any of the components of the devices used in this study;
* Concomitant use of any other eye drop;
* Concomitant use of any local or systemic treatment for dry eye;
* Concomitant use of products with known corneal toxicity and/or steroids, NSAID, or anti-glaucoma drugs;
* Concomitant hormonal therapy;
* Concomitant autoimmune inflammatory diseases or diabetes mellitus;
* Current or past participation in any other clinical trial which has ended less than a month before the enrolment;
* Use of hard contact lenses;
* Patients unlikely to cooperate in the clinical investigation or to comply with the treatment or with the clinical investigation visits.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-09-09 (Actual); Primary Completion 2022-12-18 (Actual); Study Completion 2023-11-28 (Actual)

PRIMARY OUTCOMES:
Schirmer Test | 30 days
  The test will be performed as follows:
  A standardized tear testing strips is placed between the eyeball and the lateral margin of the lower lid, the conjunctival sac of the patient, and the advancement of a tear film over a period of 5 minutes is noted. The Investigator traces the tear edge with a pen, measuring the shortest and longest parts. More than 10 mm of moisture on the filter paper after 5 minutes is a sign of normal tear production.
  Both eyes are tested at the same time and both eyes normally release the same amount of tears.
  The values obtained after 30 days of treatment will be compared with the baseline (day 0) values.
Serious Adverse Device Effects (SADE), Serious Adverse Events (SAE), Adverse Device Effects (ADE), Adverse Events (AE) and Device Deficiency (DD) | 30 days
  The occurrence of SADE, SAE, ADE, AE and DD will be monitored to assess the overall safety of the device

SECONDARY OUTCOMES:
Tear breakup time (TBUT)) | 30 days
  The test will be performed as follows:
  The fluorescein is instilled into the patient's tear film and the patient is asked not to blink while the tear film is observed under a broad beam of cobalt blue illumination. The TBUT is recorded as the number of seconds that elapse between the last blink and the appearance of the first dry spot in the tear film. A TBUT under 10 seconds is considered abnormal.
  The TBUT is able to confirm the result of the performed Schirmer test. The TBUT values obtained after 30 days of treatment will be compared with the baseline (day 0) values.
Foreign body sensation | 30 days
  The symptom will be measured using the following 4-point verbal rating scale: 0 = no symptoms; 1= mild symptoms; 2= moderate symptoms; 3= severe symptoms.
  The symptom will be collected by the patient at the time of eye drop administration and 10 minutes thereafter during the final visit (day 30)
Redness | 30 days
  The symptom will be measured using the following 4-point verbal rating scale: 0 = no symptoms; 1= mild symptoms; 2= moderate symptoms; 3= severe symptoms.
  The symptom will be collected by the patient at the time of eye drop administration and 10 minutes thereafter during the final visit (day 30)
Lachrymation | 30 days
  The symptom will be measured using the following 4-point verbal rating scale: 0 = no symptoms; 1= mild symptoms; 2= moderate symptoms; 3= severe symptoms.
  The symptom will be collected by the patient at the time of eye drop administration and 10 minutes thereafter during the final visit (day 30)
Photophobia | 30 days
  The symptom will be measured using the following 4-point verbal rating scale: 0 = no symptoms; 1= mild symptoms; 2= moderate symptoms; 3= severe symptoms.
  The symptom will be collected by the patient at the time of eye drop administration and 10 minutes thereafter during the final visit (day 30)
Discomfort | 30 days
  The symptom will be measured using the following 4-point verbal rating scale: 0 = no symptoms; 1= mild symptoms; 2= moderate symptoms; 3= severe symptoms.
  The symptom will be collected by the patient at the time of eye drop administration and 10 minutes thereafter during the final visit (day 30)
Mucus hypersecretion | 30 days
  The symptom will be measured using the following 4-point verbal rating scale: 0 = no symptoms; 1= mild symptoms; 2= moderate symptoms; 3= severe symptoms.
  The symptom will be collected by the patient at the time of eye drop administration and 10 minutes thereafter during the final visit (day 30)
Swelling | 30 days
  The symptom will be measured using the following 4-point verbal rating scale: 0 = no symptoms; 1= mild symptoms; 2= moderate symptoms; 3= severe symptoms.
  The symptom will be collected by the patient at the time of eye drop administration and 10 minutes thereafter during the final visit (day 30)
Pain/soreness | 30 days
  The symptom will be measured using the following 4-point verbal rating scale: 0 = no symptoms; 1= mild symptoms; 2= moderate symptoms; 3= severe symptoms.
  The symptom will be collected by the patient at the time of eye drop administration and 10 minutes thereafter during the final visit (day 30)
Stinging | 30 days
  The symptom will be measured using the following 4-point verbal rating scale: 0 = no symptoms; 1= mild symptoms; 2= moderate symptoms; 3= severe symptoms.
  The symptom will be collected by the patient at the time of eye drop administration and 10 minutes thereafter during the final visit (day 30)
Burning | 30 days
  The symptom will be measured using the following 4-point verbal rating scale: 0 = no symptoms; 1= mild symptoms; 2= moderate symptoms; 3= severe symptoms.
  The symptom will be collected by the patient at the time of eye drop administration and 10 minutes thereafter during the final visit (day 30)
Itching | 30 days
  The symptom will be measured using the following 4-point verbal rating scale: 0 = no symptoms; 1= mild symptoms; 2= moderate symptoms; 3= severe symptoms.
  The symptom will be collected by the patient at the time of eye drop administration and 10 minutes thereafter during the final visit (day 30)
Blurred vision | 30 days
  The symptom will be measured using the following 4-point verbal rating scale: 0 = no symptoms; 1= mild symptoms; 2= moderate symptoms; 3= severe symptoms.
  The symptom will be collected by the patient at the time of eye drop administration and 10 minutes thereafter during the final visit (day 30)
Stickiness of eyelashes | 30 days
  The symptom will be measured using the following 4-point verbal rating scale: 0 = no symptoms; 1= mild symptoms; 2= moderate symptoms; 3= severe symptoms.
  The symptom will be collected by the patient at the time of eye drop administration and 10 minutes thereafter during the final visit (day 30)
Vision changes | 30 days
  The symptom will be measured using the following 4-point verbal rating scale: 0 = no symptoms; 1= mild symptoms; 2= moderate symptoms; 3= severe symptoms.
  The symptom will be collected by the patient at the time of eye drop administration and 10 minutes thereafter during the final visit (day 30)
Discomfort on lens insertion | 30 days
  In the contact lenses wearer patients only this parameter will be evaluated (using a 4-point Verbal Rating Scale (0 = no symptoms; 1= mild symptoms; 2= moderate symptoms; 3= severe symptoms)
Discomfort on lens removal | 30 days
  In the contact lenses wearer patients only this parameter will be evaluated (using a 4-point Verbal Rating Scale (0 = no symptoms; 1= mild symptoms; 2= moderate symptoms; 3= severe symptoms)
Dryness on lens insertion | 30 days
  In the contact lenses wearer patients only this parameter will be evaluated (using a 4-point Verbal Rating Scale (0 = no symptoms; 1= mild symptoms; 2= moderate symptoms; 3= severe symptoms)
Dryness on lens removal | 30 days
  In the contact lenses wearer patients only this parameter will be evaluated (using a 4-point Verbal Rating Scale (0 = no symptoms; 1= mild symptoms; 2= moderate symptoms; 3= severe symptoms)
Stinging at 1st and 2nd hour after lens insertion | 30 days
  In the contact lenses wearer patients only this parameter will be evaluated (using a 4-point Verbal Rating Scale (0 = no symptoms; 1= mild symptoms; 2= moderate symptoms; 3= severe symptoms)
Patient General satisfaction | 30 days
  This parameter will be recorded by the patients using a 4-point Verbal Rating Scale (1= poor satisfaction, 2= moderate satisfaction; 3= good satisfaction; 4= very good satisfaction) and reported in the final visit (day 30).

CONTACTS AND LOCATIONS:
Overall Officials: Gennaro Crugliano, MD, Prof, Principal Investigator — Ospedale San Giovanni di Dio, Crotone (Italy)
Locations (1):
- USOD Oculistica, Presidio Ospedaliero di Crotone, Ospedale San Giovanni di Dio, Crotone, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] The definition and classification of dry eye disease: report of the Definition and Classification Subcommittee of the International Dry Eye WorkShop (2007). Ocul Surf. 2007 Apr;5(2):75-92. doi: 10.1016/s1542-0124(12)70081-2. PMID 17508116
- [Background] Ang BCH, Sng JJ, Wang PXH, Htoon HM, Tong LHT. Sodium Hyaluronate in the Treatment of Dry Eye Syndrome: A Systematic Review and Meta-Analysis. Sci Rep. 2017 Aug 21;7(1):9013. doi: 10.1038/s41598-017-08534-5. PMID 28827614
- [Background] Fraser JR, Laurent TC, Laurent UB. Hyaluronan: its nature, distribution, functions and turnover. J Intern Med. 1997 Jul;242(1):27-33. doi: 10.1046/j.1365-2796.1997.00170.x. PMID 9260563
- [Background] Tampucci S, Monti D, Burgalassi S, Terreni E, Zucchetti E, Baldacci F, Chetoni P. Effect of 5-Oxo-2-Pyrrolidinecarboxylic Acid (PCA) as a New Topically Applied Agent for Dry Eye Syndrome Treatment. Pharmaceutics. 2018 Aug 25;10(3):137. doi: 10.3390/pharmaceutics10030137. PMID 30149648